CLINICAL TRIAL: NCT03954782
Title: Efficacy of Nintedanib Per os as a Treatment for Epistaxis in HHT Disease. A National, Randomized, Multicentre Phase II Study
Brief Title: Efficacy of Nintedanib Per os as a Treatment for Epistaxis in HHT Disease.
Acronym: EPICURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69HCL19_0003; 2019-002593-31 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2023-08

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic; Rendu Osler Disease
Keywords: Hereditary Hemorrhagic Telangiectasia (HHT); antiangiogenic therapy; Tyrosine Kinase Inhibitor; Nintedanib
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintedanib (Experimental): Oral treatment of Nintedanib 150 mg soft capsule
  Interventions: Drug: Nintedanib 150 mg and 100 mg soft capsules
- Placebo (Placebo Comparator): Oral treatment of placebo soft capsule
  Interventions: Drug: Oral treatment of placebo soft capsule

INTERVENTIONS:
Drug: Nintedanib 150 mg and 100 mg soft capsules — Nintedanib 150 mg soft capsules twice daily approximately 12 hours apart (i.e. 300 mg/day) for 12 weeks. In case of adverse reaction a dose reduction at 200 mg/day (100 mg twice daily) can be prescribe.
  Arms: Nintedanib
Drug: Oral treatment of placebo soft capsule — Placebo soft capsules (identical to 150 mg and 100 mg soft capsules)
  Arms: Placebo

SUMMARY:
The recognized manifestations of HHT are all due to abnormalities in vascular structure. Epistaxis are spontaneous, very variable, may occur as often as several times every day, and are recurrent in 90% of patients and associated with chronic and severe anemia in 2-10%. They also significantly reduce quality of life.

Blood transfusions are sometimes required in 10-30% of patients. Previous studies showed that antiangiogenic treatments such as anti-VEGF treatment (bevacizumab) administered intravenously was efficient on epistaxis and dramatically reduced nosebleeds.

Tyrosine kinase inhibitors are anti-angiogenic molecules which are available orally and could therefore overcome the difficulties encountered with bevacizumab. The investigator hypothesized that nintedanib, acting by indirect inhibition of the VEGF receptor should allow a reduction of epistaxis in HHT patient.

Nintedanib has been used in one HHT patient following the diagnosis of Insterstitial Pulmonary Fibrosis (published case report in 2017, Kovacs et al) with encouraging results.

The aim is to evaluate efficacy of nintedanib for the treatment of epistaxis in HHT patients

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients who have given their free informed and signed consent
* Patients affiliated to a social security scheme or similar
* Patients monitored for clinically confirmed HHT and/or with molecular biology confirmation
* Patient with an Epistaxis Severity Score (ESS) > 4

Exclusion Criteria:

* Pregnant woman or woman of child bearing potential
* Woman who are breast feeding.
* Patient who is protected adults under the terms of the law (French Public Health Code).
* Participation in another interventional clinical trial which may interfere with the proposed trial
* Active infection.
* (AST, ALT > 1,5 fold upper limit of normal (ULN) and/or Bilirubin > 1,5 fold upper limit of normal (ULN).
* Severe renal impairment
* Presence of non-treated pulmonary arteriovenous malformations accessible to a treatment on CT scan within 5 years.
* Patients with hemoptysis or hematuria within 12 weeks prior to inclusion.
* Patients with active gastro-intestinal (GI) bleeding or GI ulcers within 12 months prior to inclusion.
* Presence of cerebral arteriovenous malformation.
* Patients who require full-dose therapeutic anticoagulation (e.g. vitamin K antagonist or heparin, dabigatran) or high dose antiplatelet therapy, , patients under anticoagulation with rivaroxaban, apixaban and epixaban.
* Patients with P-glycoprotein (P-gp) substrates/inducers/inhibitors (e.g.: ketoconazole, erythromycin, cyclosporine, rifampicin, carbamazepine, phenytoin, and St. John's Wort).
* Patients with known coronary artery disease or recent history of myocardial infarction (within 1 year).
* Known inherited predisposition to thrombosis or thrombotic events( including stroke and transient ischemic attack, excluded superficial venous thrombosis) within 12 months prior to inclusion.
* Patients with QTc prolongation
* Hypersensitivity to nintedanib, peanut or soya, or to any of the excipients.
* Patient who incompletely filled in epistaxis grids within 8 weeks prior to inclusion.
* Patient who have received intravenous bevacizumab within 6 months prior to inclusion.
* Patient who had surgery (including ENT (Ear, Nose and Throat Specialist) surgery) within 12 weeks prior to inclusion.
* Unhealed wound.
* Planned major surgery within the next 3 months, including liver transplantation, major abdominal or intestinal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Epistaxis duration assessed on epistaxis grids completed by the patients. | 12 weeks

SECONDARY OUTCOMES:
number of adverse events | 6 months
number of adverse events | 12 weeks
number of adverse events | 24 weeks
Efficacy or nintedanib assessed by ESS (Epistaxis Severity Score) questionnaire | 12 weeks
  This score assess the severity of epistaxis (minimum 0 corresponds to "none" and maximum 10 corresponds to"severe")
Efficacy or nintedanib assessed by ESS questionnaire | 24 weeks
  This score assess the severity of epistaxis (minimum 0 corresponds to "none" and maximum 10 corresponds to"severe")
duration of epistaxis all over the study. Assessment on epistaxis grids completed by the patients. | 12 weeks
duration of epistaxis assessed on epistaxis grids completed by the patients. | 24 weeks
duration of epistaxis assessed on epistaxis grids completed by the patients. | 12 weeks
frequency of epistaxis assessed on epistaxis grids completed by the patients. | 24 weeks
Quality of life assessed by SF36 (Short Form 36) questionnaire | 12 weeks
Quality of life assessed by SF36 questionnaire | 24 weeks
number of red blood cell transfusions | 12 weeks
number of red blood cell transfusions | 24 weeks
number of iron infusions | 12 weeks
number of iron infusions | 24 weeks
hemoglobin level | 12 weeks
hemoglobin level | 24 weeks
ferritin level | 12 weeks
ferritin level | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUPUIS-GIROD, Principal Investigator — Hospices Civils de Lyon
Locations (8):
- France (8):
  - CHU d'Angers, Angers
  - Hôpital Femme-Mère-Enfant-Centre de Référence pour la maladie de Rendu-Osler, Bron
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU de Marseille-Hôpital la conception, Marseille
  - CHU de Montpellier-Hôpital St Eloi, Montpellier
  - Hôpital Tenon, Paris
  - CHRU - Hôpital J.Bernard, Poitiers
  - CHU de Rennes-Hôpital Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hermann R, Grobost V, Le-Guillou X, Lavigne C, Parrot A, Riviere S, Seguier J, Fargeton AE, de-Montigny A, Huot M, Decullier E, Roux A, Gervaise C, Cartier C, Dufour X, Grall M, Jegoux F, Laccourreye L, Michel J, Saroul N, Wagner I, Kerjouan M, Dupuis-Girod S. Effect of oral nintedanib vs placebo on epistaxis in hereditary hemorrhagic telangiectasia: the EPICURE multicenter randomized double-blind trial. Angiogenesis. 2024 Dec 24;28(1):9. doi: 10.1007/s10456-024-09962-4. PMID 39718659